CLINICAL TRIAL: NCT06670534
Title: A Multicenter,Randomized,Open-label,Positive-controlled Study to Evaluate the Efficacy and Safety of JMKX003142 in Renal Edema Patients
Brief Title: A Dose-finding Study of JMKX003142 in Treatment of Renal Edema
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jemincare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JMKX003142-R201
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2024-10

CONDITIONS: Edema Secondary; Edema Leg
Keywords: renal edema; edema due to kidney diseases
MeSH Terms: interventions — Torsemide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- low dose group (Experimental): low dose of JMKX003142 tablets，take orally once daily，last for 7 days
  Interventions: Drug: JMKX003142 tablets
- median dose group (Experimental): median dose of JMKX003142 tablets，take orally once daily，last for 7 days
  Interventions: Drug: JMKX003142 tablets
- high dose group (Experimental): high dose of JMKX003142 tablets，take orally once daily，last for 7 days
  Interventions: Drug: JMKX003142 tablets
- active comparator group (Active Comparator): torasemide tablets 20mg，take orally once daily，last for 7 days
  Interventions: Drug: Torasemide tablets

INTERVENTIONS:
Drug: JMKX003142 tablets — JMKX003142 tablets for experimental groups.Take the JMKX003142 tablets（on empty stomach） once daily for seven days.
  Arms: high dose group; low dose group; median dose group
Drug: Torasemide tablets — Torasemide tablets for active comparator group.Take the torasemide tablets once daily for seven days.
  Arms: active comparator group

SUMMARY:
To Evaluate the Safety, Efficacy, and Pharmacokinetic Characteristics of JMKX003142 Administered Randomly, Open-label, Active-controlled Study in Chinese Renal Edema Patients.

DETAILED DESCRIPTION:
JMKX003142 is an arginine vasopressin（AVP）-V2R antagonist which shows a remarkable diuretic effect in healthy volunteers.In this phase 2 study ，we will observe the safety 、efficacy and pharmacokinetic（PK） characteristics about different dose levels of JMKX003142 tablets in renal edema patients. This phase 2 study is designed as a randomly, open-label, active-controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who can fully understand the purpose and process of the study and voluntarily sign the informed consent form（ICF）;
* Age ≥ 18 years old during screening;
* Diagnosed as renal edema during screening;
* Estimated glomerular filtration rate（eGFR） ≥ 15 mL/min/1.73m2 during screening.

Exclusion Criteria:

* Patients who are receiving the renal replacement therapy during screening or patients who require renal replacement therapy in the short term evaluated by the researchers;
* Patients who are suspected with hypovolemia;
* Patients with the following diseases or symptoms: acute thrombosis, diarrhea, and difficulty urinating;
* Patients who are unable to sense thirst or who have difficulty with fluid intake;
* Patients who have received arginine vasopressin-V2R blockers within 30 days prior to the screening examination;
* The following laboratory indicators are abnormal: glutamic pyruvic transaminase ≥ 1.5 ×upper limit of normal, glutamic oxaloacetic transaminase ≥ 1.5 × upper limit of normal, serum sodium> upper limit of normal, D-dimer ≥ 2 × upper limit of normal;
* Patients who received diuretics or treatments with diuretic effects from Day-2 to randomization;
* During screening, systolic blood pressure <90mmHg/diastolic blood pressure<60mmHg, systolic blood pressure>160mmHg/diastolic blood pressure >100mmHg;
* Patients who have a history of allergies to ≥ 3 substances, or are currently in an allergic state;
* Female patients who are breast-feeding or who have a positive pregnancy test result prior to receiving investigational product (IMP);
* Sexually active males or women of childbearing potential (WOCBP) who do not agree to practice birth control or remain abstinent during the trial and for 30 days after the final IMP administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
body weight | 7 days

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fudan University Affiliated Zhongshan Hospital, Shanghai
  - Zhejiang Hangyu Pharmaceutical Co., Ltd（subsidiary of Jemincare）, Shanghai

IPD SHARING:
Plan to Share IPD: No